CLINICAL TRIAL: NCT06488391
Title: The Impact of Patients' Daily Independent Breathing Training on the Accuracy and Side Effects of Deep Inspiratory Breath-Hold Radiotherapy for Breast Cancer
Brief Title: The Impact of Respiratory Training of DIBH Radiotherapy for Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianjun Lai (Other)
Responsible Party: Sponsor-Investigator, Jianjun Lai, Advanced Medical Physicist, Zhejiang Hospital
Organization: Zhejiang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDIBT001
Record Dates: First submitted 2024-06-21; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visualized Self-Training (Experimental)
  Interventions: Behavioral: Using a Portable Visualized Device for Self-Directed Breathing Training
- No-Visualized Self-Training (No Intervention)

INTERVENTIONS:
Behavioral: Using a Portable Visualized Device for Self-Directed Breathing Training — Using a Portable Visualized Device for Self-Directed Breathing Training
  Arms: Visualized Self-Training

SUMMARY:
Breast cancer DIBH (Deep Inspiration Breath Hold) radiotherapy represents a high-precision treatment approach that substantially minimizes radiation exposure to vital organs such as the heart, thus enhancing protection of the patient's heart, lungs, contralateral breast, and other normal tissues compared to conventional radiotherapy techniques. This method requires meticulous precision, necessitating that patients possess exceptional respiratory control, which is facilitated through specialized equipment. Without such control, patients may encounter issues like missed targets, significant setup errors, and extended treatment durations.

In this study, the research team employed portable devices to enable patients to independently perform daily respiratory training exercises. The control group received no such devices; instead, these patients were merely instructed verbally on the importance of improving their breath-holding capabilities. The effectiveness of this intervention was evaluated by comparing the daily setup errors between the two groups. Additionally, the intervention's influence on patient outcomes was assessed by monitoring the toxicity and side effects experienced by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer Radiotherapy Patients
* A single breath-hold can last for more than 10 seconds

Exclusion Criteria:

* A single breath-hold can last for more than 10 seconds

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
The daily measured setup error values of the image-guided radiotherapy device during the patient's treatment process. | 5 weeks
  Statistical comparison and analysis of daily setup error values in patients are used to evaluate the effectiveness of the intervention measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No